CLINICAL TRIAL: NCT00835718
Title: A Phase II Multicenter, Randomized, Double-Blind, Two-Stage Clinical Trial to Evaluate the Efficacy and Safety of MK0594 in Patients With Alcohol Dependence
Brief Title: A Study of MK0594 in Patients With Alcohol Dependence (0594-020)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0594-020; MK0594-020; 2009_533
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Stage I, Arm 1 (Experimental): MK0594 5 mg/day
  Interventions: Drug: Comparator: MK0594 5 mg/day
- Stage I, Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo to MK0594
- Stage II, Arm 2 (Experimental): MK0594 1 mg/day
  Interventions: Drug: Comparator: MK0594 1 mg/day
- Stage II, Arm 3 (Experimental): MK0594 1 mg/week
  Interventions: Drug: Comparator: MK0594 1 mg/week
- Stage II, Arm 4 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo to MK0594

INTERVENTIONS:
Drug: Comparator: MK0594 5 mg/day — MK0594 5 mg tablets taken orally once daily for 12 weeks. At the randomization visit, a loading dose of 15 mg MK0594 will be administered.
  Arms: Stage I, Arm 1
Drug: Comparator: MK0594 1 mg/day — MK0594 1 mg tablets taken orally once daily for 12 weeks. At the randomization visit, a loading dose of 3 mg MK0594 will be administered.
  Arms: Stage II, Arm 2
Drug: Comparator: MK0594 1 mg/week — MK0594 1 mg tablets taken orally once every 7 days for 12 weeks. At the randomization visit, a loading dose of 3 mg MK0594 will be administered.
  Arms: Stage II, Arm 3
Drug: Comparator: Placebo to MK0594 — Matching placebo to MK0594 tablets taken orally once daily for 12 weeks.
  Arms: Stage I, Arm 2; Stage II, Arm 4

SUMMARY:
A study in patients with alcohol dependence to see if MK0594 is safe and effective in maintaining absence of heavy drinking over a 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patient has Diagnostic and Statistical Manual of Mental Disorders, fourth edition, text revision diagnosis of alcohol dependence and alcohol addiction
* Patient has two heavy drinking days in the last 30 days
* Patient has 3 days of abstinence from alcohol right before taking study medication
* Patient has lived in the same residence for the last 2 months

Exclusion Criteria:

* If female, patient is pregnant or breastfeeding
* Patient anticipated inpatient alcohol treatment
* Patient has a history of suicide attempt in the last year
* Patient has schizophrenia or bipolar disorder
* Patient has a history of multiple or serious allergies
* Patient has participated in a clinical trial in the last 30 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-02-27 (Actual); Primary Completion 2010-03-11 (Actual); Study Completion 2010-03-11 (Actual)

PRIMARY OUTCOMES:
no heavy alcohol drinking and safety as measured by adverse experiences, laboratory safety test, vital signs, ECG, and physical examination | week 3 and 12 after starting study medication for efficacy and over 12 weeks and 52 weeks for safety
  no heavy alcohol drinking and safety as measured by adverse experiences, laboratory safety test, vital signs, ECG, and physical examination

SECONDARY OUTCOMES:
no alcohol drinking | week 3 to 12 after starting study medication and over 52 weeks
  no alcohol drinking

CONTACTS AND LOCATIONS:
Overall Officials: Menlo Therapeutics Inc., Study Director — Vyne Therapeutics Inc.